CLINICAL TRIAL: NCT03715010
Title: Effects of Branch Chain Amino Acids on Glucose Tolerance in Obese Pre-diabetic Subjects
Brief Title: Investigation of an Amino Acid Supplement on Glucose Levels in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-001928
Record Dates: First submitted 2018-10-09; First posted 2018-10-22 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Pre-diabetes; Obese; Glucose Intolerance
MeSH Terms: conditions — Glucose Intolerance; Obesity | interventions — Amino Acids

STUDY DESIGN:
Intervention Model Description: BCAA
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain Chain Amino Acid (BCAA) (Active Comparator): Subjects will be randomly assigned to take either the 25g supplement (containing 4g BCAA) daily for 4 weeks followed by the 20g BCAA supplement daily for 4 weeks, or vice versa, cross-over design
  Interventions: Dietary Supplement: BCAA
- Placebo (Placebo Comparator): Subjects will be randomly assigned to take either the 25g supplement (containing 4g BCAA) daily for 4 weeks followed by the 20g BCAA supplement daily for 4 weeks, or vice versa, cross-over design
  Interventions: Dietary Supplement: BCAA

INTERVENTIONS:
Dietary Supplement: BCAA — Subjects will be randomly assigned to take either the 25g supplement (containing 4g BCAA) daily for 4 weeks followed by the 20g BCAA supplement daily for 4 weeks, or vice versa
  Other Names: Branch Chain Amino Acid

SUMMARY:
This study aims to determine whether the use of Branched-Chain Amino Acids (BCAA's) regulate insulin and glucagon secretion, and whether the supplement has any effect on body weight and body composition. Subjects who participate in this study will receive an 8-week supply of supplement. The study supplements will be manufactured by Scientific Living, in Irvine, CA for high dose BCAA and the low dose BCAA is manufactured by Nutribiotic, Lakeport, CA. Timed blood collections will be used to measure how BCAA affect glucose metabolism/insulin sensitivity in human subjects.

DETAILED DESCRIPTION:
1. BCAA's multiple functions in cells In addition to participating in de novo protein synthesis, Branched-Chain Amino Acids (BCAAs, including leucine, isoleucine, and valine) regulate multiple cellular functions as nutrient signaling. For example, BCAAs regulate insulin and glucagon secretion and thus glucose metabolism1. BCAAs, especially leucine, is one key regulator of mTOR signaling, which is the central component of a complex signaling network of insulin signaling, cell growth, and proliferation. BCAAs also regulate protein synthesis and degradation in various tissues.
2. Impact of BCAA supplemental or BCAA-enriched diet on metabolism In addition to the healthcare utilization of BCAAs for liver disorders and their complications and other diseases, BCAA supplementation is common amongst athletes and fitness professionals to improve muscle building and strength. Meanwhile, BCAA supplementation or BCAA-rich protein diets are often associated with positive effects on body weight and glucose homeostasis1. Increasing dietary uptake of BCAAs improved the parameters associated with obesity and T2DM, such as body composition and glycemia levels. However, these beneficial effects are not conclusive. Moreover, other studies have shown that circulating branched-chain amino acid concentrations are associated with obesity and future insulin resistance in children and adolescents2.
3. Summary Both beneficial and detrimental effects of BCAA on metabolism have been established and therefore warrants further investigation. In the preliminary study, we found that BCAAs enhanced glucose metabolism in lean mice while they promoted glucose intolerance in obese mice. In lean mice, BCAAs decreased adiposity and enhanced glucose utilization and insulin sensitivity in different tissues. But in obese mice, BCAAs' effects were mediated by impaired insulin signaling in fat tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-65 years of age at screen
2. BMI between 27 to 40
3. Fasting glucose level >100, but <126 mg/dL or HgbA1c >5.7% but < 6.4%
4. Waist circumference > 40 in for men and >35 in for women
5. Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent.

Exclusion Criteria:

1. Any subject with a history of diabetes mellitus on medications, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, cancer (except skin basal cell carcinoma ) chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP>160mmHg, diastolic BP>95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
2. Any subject with a screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
3. Any subject who currently uses tobacco products.
4. Any history of gastrointestinal disease except for appendectomy.
5. Any antibiotic or laxative use during the 2 months before the study.
6. Any subject who is unable or unwilling to comply with the study protocol.
7. Any subject allergic to soy products.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-03-18 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Measure of glucose AUC during 2H OGTT (Frame: 10 weeks) | Baseline week4, week6 and 10 weeks
  To assess change of glucose AUC during 2H OGTT test

SECONDARY OUTCOMES:
Measure of body composition (Time Frame: 10 weeks) | Baseline week4, week6 and 10 weeks
  To assess changes in body composition (fat mass, lean body mass in Kg)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutriiton, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woo SL, Yang J, Hsu M, Yang A, Zhang L, Lee RP, Gilbuena I, Thames G, Huang J, Rasmussen A, Carpenter CL, Henning SM, Heber D, Wang Y, Li Z. Effects of branched-chain amino acids on glucose metabolism in obese, prediabetic men and women: a randomized, crossover study. Am J Clin Nutr. 2019 Jun 1;109(6):1569-1577. doi: 10.1093/ajcn/nqz024. PMID 31005973